CLINICAL TRIAL: NCT00003585
Title: A Phase I/II Pilot Study of a Novel Four Drug Regimen for the Treatment of Advanced Renal Cell Carcinoma: FUNIL-cRA
Brief Title: Biological Therapy Plus Chemotherapy in Treating Patients With Metastatic or Recurrent Kidney Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: UNM-0996C; CDR0000066654 (Registry Identifier: PDQ (Physician Data Query)); NCI-V98-1478
Record Dates: First submitted 1999-11-01; First posted 2004-07-22 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Kidney Cancer
Keywords: stage IV renal cell cancer; recurrent renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — aldesleukin; Interferon-alpha; Fluorouracil; Isotretinoin; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: aldesleukin
Biological: recombinant interferon alfa
Drug: fluorouracil
Drug: isotretinoin
Procedure: surgical procedure

SUMMARY:
RATIONALE: Biological therapies use different ways to stimulate the immune system and stop cancer cells from growing. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining biological therapy with chemotherapy may kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of biological therapy plus chemotherapy in treating patients with metastatic or recurrent kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the toxic effects, patient tolerance, and practicality of administering interferon alfa-2b, fluorouracil, interleukin-2, and isotretinoin (FUNIL-cRa) in patients with metastatic and/or recurrent renal cell carcinoma. II. Obtain a pilot indication of responsiveness of these patients to this regimen. III. Evaluate the measurement of tumor thymidylate synthetase as a prediction of response of these patients to this and other fluorouracil based regimens.

OUTLINE: Patients are stratified by performance status (0 vs 1), nephrectomy (yes vs no), site of disease (pulmonary or lymph node metastases only vs other disease site), radiotherapy (yes vs no), and prior adjuvant biologic or hormone therapy (yes vs no). Patients receive intravenous fluorouracil daily for 14 days, and subcutaneous interferon alfa-2b 3 times a week for 6 weeks. Beginning on day 15, patients receive intravenous interleukin-2, 5 days a week and oral isotretinoin 2 times a day for 4 weeks. Treatment courses are 6 weeks, followed by a 2 week rest period. Treatment continues for up to 4 courses in the absence of disease progression or unacceptable toxicity. Patients with partial or complete response may undergo surgical resection. Patients are followed every 2 months for 1 year and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 35 patients will be accrued to this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven metastatic and/or recurrent renal cell carcinoma Bidimensionally measurable disease No concurrent brain metastases Patients with prior brain metastases who have undergone radiation and/or surgery, with stable response, confirmed by MRI, and off corticosteroids are eligible

PATIENT CHARACTERISTICS: Age: Not specified Performance status: SWOG 0-1 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: Not pregnant or nursing Fertile patients must use effective contraception No other serious illness or active infection requiring antibiotics Not HIV positive No active substance abuse

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 6 months since prior interleukin-2 therapy At least 6 months since prior interferon alfa therapy At least 1 month since other prior biologic therapy No other concurrent biologic therapy (e.g., filgrastim or sargramostim) Chemotherapy: At least 6 months since prior fluorouracil therapy At least 1 month since prior chemotherapy No other concurrent chemotherapy Endocrine therapy: At least 1 month since prior endocrine therapy No concurrent hormone therapy No concurrent corticosteroids except if inhaled or topical Radiotherapy: At least 1 month since prior radiotherapy (to less than 25% of the bone marrow only, and there must be measurable disease outside of radiation field) No concurrent radiotherapy Surgery: At least 3 weeks since prior surgery Other: No concurrent ongoing therapy with investigational drugs

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 1996-08; Primary Completion 2001-08 (Actual); Study Completion 2002-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Elias, MD, Study Chair — University of New Mexico Cancer Center
Locations (1):
- University of New Mexico Cancer Research & Treatment Center, Albuquerque, New Mexico, United States